CLINICAL TRIAL: NCT04117490
Title: A Double Blind, Double Dummy, Dose Response, Randomized, Placebo Controlled Study to Assess the Efficacy of Epiitalis on Knee Pain in Patients Suffering From Knee Osteoarthritis
Brief Title: To Assess Efficacy of Epiitalis on Knee Pain in Patients Suffering From Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vedic Lifesciences Pvt. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: IP/190401/EPIITALIS/OA
Record Dates: First submitted 2019-10-03; First posted 2019-10-07 (Actual); Last update posted 2022-02-01 (Actual); Status verified 2020-11

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Epiitalis low dose (Active Comparator): Two capsules twice daily 30 mins before meals (breakfast & dinner).
  Interventions: Other: Epiitalis
- Epiitalis mid dose (Active Comparator): Two capsules twice daily 30 mins before meals (breakfast & dinner).
  Interventions: Other: Epiitalis
- Epiitalis high dose (Active Comparator): Two capsules twice daily 30 mins before meals (breakfast & dinner).
  Interventions: Other: Epiitalis
- Placebo (Placebo Comparator): Two capsules twice daily 30 mins before meals (breakfast & dinner).
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Epiitalis — Two capsules twice daily 30 mins before meals (breakfast & dinner).
  Arms: Epiitalis high dose; Epiitalis low dose; Epiitalis mid dose
Other: Placebo — Two capsules twice daily 30 mins before meals (breakfast & dinner).
  Arms: Placebo

SUMMARY:
Epiitalis is an ingredient of a currently marketed product named as Osteo-Restore, indicated for joint health.The present study is primarily planned to establish the role of Epiitalis as a single ingredient in the treatment of mild to moderate cases of knee Osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

1. Male & female aged ≥ 40 to ≤ 65 years suffering from primary idiopathic osteoarthritis of the knee diagnosed at least 3 months prior to screening.

2 BMI ≥ 18 and ≤ 29.9 kg/m2. 3 Fasting blood sugar ≤ 126 mg/dl 4 LFT: Serum Glutamic oxaloacetic transaminase (SGOT) & <2X Upper Limit of Normal (UNL) and Serum Glutamic-Pyruvic transaminase (SGPT) & <2X UNL.

5 Serum Creatinine & <1.5X UNL. 6 Index knee joint pain rated ≥ 60 on a 100-point Pain-Visual Analogue Scale (VAS).

7. Osteoarthritis grade II/ III (Kellgren-Lawrence classification) as confirmed by: Grade II - Definite osteophytes and possible joint space narrowing (JSN) on the anteroposterior weight-bearing radiograph Grade III - Multiple osteophytes, definite JSN, sclerosis, and possible bony deformity 8. Systolic blood pressure & <140 mmHg and diastolic blood pressure & < 90 mmHg 9. In the case of hypothyroidism, only euthyroid patients will be allowed to be screened further. Blood reports of last 3 months will be valid at the time of screening.

10. Female participants of childbearing age must be willing to use the accepted methods of contraception during the course of the study.

11. Participants should be willing to be involved in some

Exclusion Criteria:

1. History of osteoarthritis for more than 3 years.
2. History of osteoporosis and/or frequent fractures.
3. History of major trauma to the index joint.
4. History of arthroscopic surgery or intervention on the index joint or awaiting a replacement of knee or hip joint.
5. History of restless leg syndrome.
6. Participants who have received intra-articular steroids or hyaluronic acid within the last three months.
7. Not willing to abstain from the use of NSAIDs (including low dose aspirin 50 mg/day for cardiovascular health) or herbal/ nutraceutical supplements for joint health.
8. Not willing to abstain from application of local analgesics, herbal oil 48 hours prior to study visit.
9. Use of any immunosuppressive drugs in the last 12 months (including steroids).
10. Participants with deformity of the knee joint.
11. Participants categorized as ACR Functional Class I osteoarthritis
12. Participants who are significantly incapacitated or disabled and would be categorized as ACR Functional Class IV osteoarthritis (largely or wholly incapacitated), or unable to walk without assistive devices.
13. Participants with other known rheumatic or inflammatory diseases such as rheumatoid arthritis, osteomyelitis, and bone metastasis.
14. Current smokers or chronic alcoholics.
15. History of bleeding disorders.
16. Participants suffering from deep vein thrombosis.
17. Participants suffering from diabetic neuropathy.
18. History of major chronic hepatic, cardiovascular, neurological or immunosuppressive conditions or the presence of any infections.
19. Participants planning to travel in the next 56 days or engage in any non-routine activity that is likely to strain the knees.
20. Participants having a history of any malignancy.
21. Inability to comply with the protocol requirements.
22. Participation in any other clinical trial within 3 months of registering in this trial.
23. . Women of child-bearing potential with a positive pregnancy test or who are lactating.
24. Any other condition which in the opinion of the Investigator may jeopardize the study.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 237 (Actual)
Dates: Start 2019-12-12 (Actual); Primary Completion 2020-10-21 (Actual); Study Completion 2020-10-21 (Actual)

PRIMARY OUTCOMES:
Effect of consumption of IP on knee joint pain as assessed by the change in the 100-point Visual Analogue Scale (VAS) from baseline and when compared with the placebo. | From baseline to 56 days
  Participant's assessment of pain will be done on a 100 mm Visual Analogue Scale (Pain), where 0 means no pain and 100 means unbearable pain.

SECONDARY OUTCOMES:
Quality of life as assessed by a SF-36 questionnaire | From baseline to 56 days
  The 36 Item Short Form Health Survey (SF36) Questionnaire is a set of generic, coherent, and easily administered quality of life measures. These measures rely upon participant self reporting.
Effect of IP consumption and the placebo on Knee joint pain, Knee joint stiffness & Knee joint function as assessed by a specific questionnaire | From baseline to 56 days
  WOMAC is a widely used questionnaire for Osteoarthritis. WOMAC Index is a tri dimensional self administered questionnaire to assess joint pain, stiffness & physical function. WOMAC Pain comprises of 5 questions related to knee joint pain that score fro 0 to 4 (0 means no pain & 4 means extreme pain). WOMAC Stiffness consists of 2 items (score 0-4, 0 means no stiffness and 4 means extreme stiffness). WOMAC Physical function consists of 17 items with scores 0 to 4 with same scoring pattern.

CONTACTS AND LOCATIONS:
Locations (8):
- India (8):
  - Kurla Nursing Home, Mumbai, Maharashtra
  - Sai Baba Hospital, Mumbai, Maharashtra
  - Diamond Hospital, Mumbai, Maharashtra
  - Ayush Nursing Home, Mumbai, Maharashtra
  - Dinanath Orthopaedic Nursing Home, Mumbai, Maharashtra
  - K. K. Medical Centre, Mumbai, Maharashtra
  - Healthcare Medical Center and diagnostics, Mumbai, Maharashtra
  - Rainbow multispeciality hospital and trauma center, Navi Mumbai, Maharashtra

REFERENCES:
- [Derived] Mitchell PG, Bright CA, Bright DR, Srivastava SN, Raote SS, Kumar S. The Biota orientalis, oil extract Epiitalis(R), is efficacious at reducing the symptoms of knee osteoarthritis: a pilot, multi-site, dose-ranging, randomized, blinded, placebo-controlled trial. Inflammopharmacology. 2022 Aug;30(4):1323-1334. doi: 10.1007/s10787-022-01013-y. Epub 2022 Jun 22. PMID 35732989